CLINICAL TRIAL: NCT00641524
Title: Evaluation of Phlebotomy as a Treatment for Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: beatonclf
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver disease; liver fibrosis; metabolic syndrome; iron overload; phlebotomy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Metabolic Syndrome; Iron Overload | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Other): Iron depletion via phlebotomy
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Phlebotomy involves the removal of blood (approximately 500mL) each week until body iron levels reach the low-normal level
  Other Names: Venesection

SUMMARY:
The purpose of this study is to evaluate the use of phlebotomy (blood taking)as a treatment for patients with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
In this study phlebotomy will be evaluated as a therapy for non-alcoholic fatty liver disease (NAFLD), a common and important cause of liver disease. Phlebotomy has been used for many years in the treatment of disorders of iron overload such as hemochromatosis, where it is well tolerated and improves symptoms and survival. There is some evidence that it is also effective in treating NAFLD. However, previous studies have not evaluated whether phlebotomy improves liver biopsy findings. We will measure the severity disease in NAFLD patients prior to phlebotomy therapy and again at the end of treatment. This will allow us to accurately determine the benefit of this therapy in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18y or older
* Diagnosis of Non-alcoholic Fatty Liver Disease

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Alcohol consumption of >10g/day for women and >20g/day for men

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Severity of liver disease | 6 months after final treatment

SECONDARY OUTCOMES:
Severity of metabolic disease | 6 months after final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melanie D Beaton, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Beaton MD, Chakrabarti S, Levstik M, Speechley M, Marotta P, Adams P. Phase II clinical trial of phlebotomy for non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2013 Apr;37(7):720-9. doi: 10.1111/apt.12255. Epub 2013 Feb 26. PMID 23441892